CLINICAL TRIAL: NCT03796494
Title: Behavior of the Peri-implant Tissues on the Multiposition Abutment Straight Aesthetic Slim Anti-rotational Galimplant
Brief Title: Peri-implant Tissues on Aesthetic Slim Abutment Galimplant (PSG)
Acronym: (PSG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Galimplant Dental Implants (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor Mario Perez Sayans MD, PhD (Principal investigator), University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-2019-01
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2020-03

CONDITIONS: Dental Implant Failed; Dental Prosthesis Failure
Keywords: dental implant; periimplant tissues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The control group is considered, using the company's classic multi-position straight anti-rotational abutment
  Interventions: Procedure: Straight abutment
- Test group (Experimental): The test group is considered, where the new multi-position straight esthetic anti-rotational slim abutment is used
  Interventions: Procedure: Slim abutment

INTERVENTIONS:
Procedure: Straight abutment — This is the classic abutment, straight and anti-rotational for dental implants which have been tested before
  Arms: Control Group
Procedure: Slim abutment — This is the new concept of the prostheses abutment, slim and anti-rotational to improve the width of biologic space
  Arms: Test group

SUMMARY:
This is a randomized, single-blind, split-mouth clinical trial to evaluate the performance of peri-implant tissues (bone and soft tissues) in conventionally loaded Galimplant implants, using a classic multi-position, anti-rotational abutment, comparing it to the new multi-abutment aesthetic slim anti-rotational placed both at the time of the implant surgery. To this end, 80 Galimplant implants with a diameter of 4 mm and 10 mm in length will be placed in areas of mature scarred post-extraction bone. Patients be divided into 2 study groups, group C: straight pillar; Group T: Slim pillar. The bone and clinical radiological stability of the peri-implant tissues will be evaluated at 6 weeks post-surgery and at 6-12-24 months post-prosthetic loading.

ELIGIBILITY:
Inclusion Criteria:

* Patients without systemic pathology that are grounds for absolute contraindication
* Older adults who agree to be part of the study and sign the informed consent
* Consumption of tobacco less than 5 cigarettes / day
* Do not be completely toothless
* Absences of at least two pieces in posterior area with or without free ends to distal, maxillary or mandibular that do not require regenerative techniques. In case of odd absences (3,5,7), a Slim pillar will be placed, being the group to always be the majority.
* Area of mature bone healed at least 6 months post-extraction.
* Patients with a sufficient amount of bone to place implants 4 mm in diameter and 10 mm long

Exclusion Criteria:

* Immunosuppressed
* Aesthetic edentulous areas of 13-23 and 33-43
* Smokers of more than 5 cigarettes
* Index of bleeding greater than 30%
* Patients with less than 2 mm of keratinized gingiva
* Implants with primary stability with ISQ <55
* Implants with ISQ index <55 at 8 weeks
* When a margin of safety can not be assumed to the inferior dental nerve of at least 1 mm

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Primary stability of implants and peri-implant tissues | 10 months
  Randomly and following the inclusion and exclusion criteria, the implants will be placed with the normal preparation protocol. Investigators will evaluate the immediate post-surgical stability of implants and peri-implant tissues through the Ostell system, based on the resonance frequency analysis (RFA). The implant stability quotient (ISQ) is the value on a scale that indicates the level of stability and osseointegration in dental implants. The scale ranges from 1 to 100, with higher values indicating greater stability. The acceptable stability range lies between 55-85 ISQ

SECONDARY OUTCOMES:
Basal Peri-implant tissue level: implant stability | 1 day
  Randomly and following the inclusion and exclusion criteria, the implants will be placed with the normal preparation protocol. We will load the crowns 8 weeks after implant surgery. Investigators will evaluate the stability at different moments, 8 weeks, 6 months, 12 months and 24 months. The implant stability quotient (ISQ) is the value on a scale that indicates the level of stability and osseointegration in dental implants. The scale ranges from 1 to 100, with higher values indicating greater stability. The acceptable stability range lies between 55-85 ISQ. ISQ values are obtained using resonance frequency analysis (RFA).
Basal Radiological Bone Implant level | 1 day
  At the moment of placing the implant, clinical variables will be evaluated: depth of probing (distance from the peri-implant margin to the most depth of the peri-implant sulcus). This will be the basal measure of the implant stability and peri-implant tissue levels. Investigators will calculate the difference between the basal measure and the future measurements.
Basal Peri-implant tissue level: probing depth | 1 day
  At the moment of placing the implant, clinical variables will be evaluated: depth of probing (distance from the peri-implant margin to the most depth of the peri-implant sulcus). This will be the basal measure of the implant stability and peri-implant tissue levels. Investigators will calculate the difference between the basal measure and the future measurements.
Radiological bone implant stability | 8 weeks
  After the implantation, we´ll load the temporary 8 weeks after the implantation. Investigators will evaluate the bone level stability at 6 weeks in both groups, through a dental X-ray radiography. The bone stability will be measured as a difference between de basal bone level and the actual one in mm.
Peri-implant tissue stability: probing depth | 8 weeks
  After the implantation, we´ll load the definitive prostheses in 8 weeks. Investigators will evaluate the peri-implant tissue stability by measuring the probing depth or just in case, the recession of the gingival margin. The stability will be given by the differences between both measures, basal and actual in mm.
Peri-implant tissue stability: ISQ | 8 weeks
  After the implantation, we´ll load the temporary prostheses in 8 weeks. Investigators will evaluate the peri-implant tissue stability by measuring the ISQ through RFA. The stability will be given by the differences between both measures, basal and actual.

OTHER OUTCOMES:
6-months clinical evaluation of probing depth | 6 months
  After 6 months of loading of final ceramic restoration, investigators will evaluate the differences of clinical (mm of probing depth) aspects.
6-months ISQ evaluation | 6 months
  After 6 months of loading of final ceramic restoration, investigators will evaluate the differences of ISQ implant stability aspects.
  ISQ, or Implant Stability Quotient, is a scale from 1 to 99 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
6-months radiological evaluation of definitive prostheses | 6 months
  After 6 months of loading of final ceramic restoration, investigators will evaluate the differences of radiological aspects (bone implant level in mm calculated from the neck to the actual bone level), comparing on the basal and final values.
Long-term Radiological bone implant stability | 24 months
  After 24 months of loading of final ceramic restoration, investigators will evaluate the bone level stability at 24 months in both groups, through a dental X-ray radiography. The bone stability will be measured as a difference between de basal bone level and the actual one in mm.
Long-term Peri-implant tissue stability: ISQ | 24 months
  After 24 months of loading of final ceramic restoration, investigators will evaluate the peri-implant tissue stability by measuring the ISQ through Resonance Frequency Analysis (RFA). ISQ, or Implant Stability Quotient, is a scale from 1 to 99 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
  The stability will be given by the differences between both measures, basal and actual.
Long-term Peri-implant tissue stability: probing depth | 24 months
  After 24 months of loading of final ceramic restoration, investigators will evaluate the peri-implant tissue stability by measuring the probing depth or just in case, the recession of the gingival margin. The stability will be given by the differences between both measures, basal and actual in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Pérez Sayáns, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will anonymize and categorize the clinical and radiological data of the patients to share the information with the other researchers of the group
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Time Frame:
Access Criteria: under request

REFERENCES:
- See also: GI-1319 — http://imaisd.usc.es/grupoficha.asp?idpersoatipogrupo=75189&i=es&s=-2-26-148